CLINICAL TRIAL: NCT05952869
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-0616 in Adults With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study of Enlicitide Decanoate (MK-0616 Oral PCSK9 Inhibitor) in Adults With Heterozygous Familial Hypercholesterolemia (MK-0616-017) CORALreef HeFH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0616-017; MK-0616-017 (Other: MSD); 2022-502782-14-00 (Registry Identifier: EU CT); U1111-1285-4257 (Registry Identifier: UTN)
Record Dates: First submitted 2023-07-10; First posted 2023-07-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Decanoate (Experimental): Participants will receive 20 mg of enlicitide decanoate orally once daily (QD) for up to 52 weeks.
  Interventions: Drug: Enlicitide Decanoate
- Placebo (Placebo Comparator): Participants will receive enlicitide decanoate-matching placebo orally QD for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enlicitide Decanoate — Oral tablet
  Other Names: MK-0616
  Arms: Enlicitide Decanoate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the efficacy, safety, and tolerability of enlicitide decanoate in adult participants with heterozygous familial hypercholesterolemia. The primary hypothesis is that enlicitide decanoate is superior to placebo on mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Has possible or definite diagnosis of heterozygous familial hypercholesterolemia (HeFH) based on a locally accepted diagnostic algorithm
* Has an LDL-C ≥55 mg/dL or ≥70 mg/dL depending on medical history
* Is treated with a moderate- or high-intensity statin medication
* Is on a stable dose of all background lipid-lowering therapies (LLTs) with no planned medication change

Exclusion Criteria:

* Has a history of homozygous familial hypercholesterolemia (FH) based on genetic or clinical criteria, compound heterozygous FH, or double heterozygous FH
* Has a history of heart failure or heart failure hospitalization within 3 months before first study visit
* Is undergoing or previously underwent an LDL-C apheresis program within 3 months before first study visit or plans to initiate an LDL-C apheresis program
* Was previously treated/is being treated with certain other cholesterol lowering medications, including protein convertase subtilisin/kexin type 9 (PCSK9) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in LDL-C.
Number of participants with one or more adverse events (AEs) | Up to ~60 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study drug due to an AE | Up to ~52 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Mean percent change from baseline in LDL-C at Week 52 | Baseline and Week 52
  Blood samples will be collected at baseline and at Week 52 to assess mean percent change in LDL-C.
Mean percent change from baseline in non-high-density lipoprotein cholesterol (HDL-C) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in non-HDL-C.
Mean percent change from baseline in apolipoprotein B (ApoB) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess mean percent change in ApoB.
Percent change from baseline in lipoprotein(a) (Lp[a]) at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess percent change in Lp(a).
Percentage of participants with LDL-C <70 mg/dL and ≥50% reduction from baseline at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess the percentage of participants who have LDL-C <70 mg/dL and ≥50% reduction from baseline.
Percentage of participants with LDL-C <55 mg/dL and ≥50% reduction from baseline at Week 24 | Baseline and Week 24
  Blood samples will be collected at baseline and at Week 24 to assess the percentage of participants who have LDL-C <55 mg/dL and ≥50% reduction from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (59):
- United States (13):
  - Alliance for Multispecialty Research, LLC ( Site 0023), Daphne, Alabama
  - Excel Medical Clinical Trials ( Site 0008), Boca Raton, Florida
  - Advanced Pharma Research ( Site 0007), Cutler Bay, Florida
  - Progressive Medical Research ( Site 0021), Port Orange, Florida
  - Clinical Site Partners LLC, dba CSP Orlando ( Site 0028), Winter Park, Florida
  - Synexus Clinical Research US - Evansville ( Site 0031), Evansville, Indiana
  - Franciscan Physician Network - Indiana Heart Physicians ( Site 0040), Indianapolis, Indiana
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0001), Troy, Michigan
  - Velocity Clinical Research at The Pioneer Heart Institute, Lincoln ( Site 0026), Lincoln, Nebraska
  - Jubilee Clinical Research ( Site 0030), Las Vegas, Nevada
  - Wake Forest Baptist Health-Cardiovascular Medicine ( Site 0041), Winston-Salem, North Carolina
  - Velocity Clinical Research, Salt Lake City ( Site 0004), West Jordan, Utah
  - Health Research of Hampton Roads, Inc. ( Site 0020), Newport News, Virginia
- Australia (2):
  - Royal Prince Alfred Hospital-6West CV Ambulatory Care ( Site 2808), Camperdown, New South Wales
  - Victorian Heart Hospital-Monash Cardiovascular Research Centre (MCRC) ( Site 2803), Clayton, Victoria
- Brazil (3):
  - Universidade Federal Do Ceara ( Site 0702), Fortaleza, Ceará
  - Instituto Dante Pazzanese de Cardiology-Fundação Adib Jatene ( Site 0701), São Paulo, São Paulo
  - Incor - Instituto do Coracao ( Site 0703), São Paulo
- Canada (3):
  - Ecogene-21 ( Site 0510), Chicoutimi, Quebec
  - Institut de Cardiologie de Montreal ( Site 0506), Montreal, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0513), Trois-Rivières, Quebec
- Chile (4):
  - Clinical Research Chile SpA ( Site 0804), Valdivia, Los Ríos Region
  - CDIEM ( Site 0814), Providencia, Region M. de Santiago
  - Enroll SpA ( Site 0803), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-CICUC ( Site 0812), Santiago, Region M. de Santiago
- Colombia (4):
  - Fundación Centro de Investigación Clínica CIC ( Site 0906), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0903), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 0902), Barranquilla, Atlántico
  - Salud SURA Calle 100 ( Site 0918), Bogotá, Cundinamarca
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice-Interni kardiologicka klinika ( Site 3602), Brno, Brno-mesto
  - Institut Klinicke a Experimentalni Mediciny ( Site 3601), Prague, Praha 4
  - Fakultni Nemocnice u sv. Anny v Brne ( Site 3604), Brno, South Moravian
- Meilahden tornisairaala - Meilahti Tower Hospital ( Site 1300), Helsinki, Uusimaa, Finland
- Hong Kong (2):
  - Queen Mary Hospital-Medical ( Site 3300), Pok Fu Lam
  - Prince of Wales Hospital ( Site 3304), Shatin
- Hungary (3):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Belgyógyászati Klinika ( Site 1603), Szeged, Csongrád megye
  - Semmelweis Egyetem-Városmajori Szív- és Érgyógyászati Klinika ( Site 1600), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Anyagcsere Tanszék) ( Site 1601), Debrecen
- Israel (4):
  - Shaare Zedek Medical Center ( Site 1710), Jerusalem
  - Hadassah Medical Center ( Site 1709), Jerusalem
  - Rabin Medical Center ( Site 1717), Petah Tikva
  - Clalit Health Services - Sakhnin Community Clinic-Research Unit ( Site 1700), Sakhnin
- Netherlands (4):
  - Radboudumc-internal medicine ( Site 1952), Nijmegen, Gelderland
  - Amsterdam UMC, locatie AMC-Vascular Medicine Clin Trial Unit ( Site 1954), Amsterdam, North Holland
  - Vasculair Onderzoek Centrum Hoorn ( Site 1953), Hoorn, North Holland
  - Universitair Medisch Centrum Utrecht-Vascular Medicine Research ( Site 1955), Utrecht
- New Zealand (2):
  - Pacific Clinical Research Network - Rotorua ( Site 2902), Rotorua, Bay of Plenty
  - New Zealand Clinical Research (Christchurch) ( Site 2901), Christchurch, Canterbury
- Norway (2):
  - Nordlandssykehuset ( Site 2001), Bodø, Nordland
  - Oslo Universitetssykehus Aker-Lipidklinikken ( Site 2000), Oslo
- Singapore (2):
  - National University Hospital-Department of Medicine ( Site 3212), Singapore, Central Singapore
  - Changi General Hospital ( Site 3211), Singapore, Central Singapore
- Spain (3):
  - Hospital de Sant Joan Despí Moisès Broggi ( Site 2335), Sant Joan Despí, Catalonia
  - SALUT SANT JOAN DE REUS-BAIX CAMP (EDP)-Vascular and Metabolism Unit ( Site 2329), Reus, Tarragona
  - HOSPITAL CLINICO DE VALENCIA ( Site 2321), Valencia, Valenciana, Comunitat
- Taiwan (4):
  - Mackay Memorial Hospital -Tamshui Branch ( Site 3109), New Taipei City, New Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital ( Site 3106), Taipei City, Taipei
  - National Cheng Kung University Hospital-Internal Medicine ( Site 3107), Tainan
  - National Taiwan University Hospital ( Site 3100), Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Ballantyne CM, Gellis L, Tardif JC, Banka P, Navar AM, Asprusten EA, Scott R, Stroes ESG, Froman S, Mendizabal G, Wang F, Catapano AL. Efficacy and Safety of Oral PCSK9 Inhibitor Enlicitide in Adults With Heterozygous Familial Hypercholesterolemia: A Randomized Clinical Trial. JAMA. 2026 Jan 13;335(2):129-139. doi: 10.1001/jama.2025.20620. PMID 41206969
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26188&tenant=MT_MSD_9011